CLINICAL TRIAL: NCT00497887
Title: Observational Study for Identification of Genetic- and Biological-Markers of Predisposition to Atherosclerosis: Leipzig-Heart Study (LE-Heart)
Brief Title: Genetic- and Biological-Markers of Predisposition to Atherosclerosis: Leipzig-Heart Study
Acronym: LE-Heart
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Joachim Thiery, Daniel Teupser, Stephan Gielen, Gerhard Schuler, University Leipzig
Other Study IDs: 276-2005
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-01

CONDITIONS: Atherosclerosis; Coronary Arteriosclerosis; Carotid Artery Diseases; Genetic Predisposition to Disease; Biological Markers
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Carotid Artery Diseases; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, whole blood (DNA), blood cells
Oversight: Data Monitoring Committee: No

SUMMARY:
Atherosclerotic cardiovascular disease is the major cause of morbidity and mortality in Western societies. It is a complex genetic disorder with many genes involved and significant gene-environment interactions. The aim of the study is to identify novel genetic- and biological-markers of atherosclerosis. Atherosclerosis is assessed in the coronary arteries using coronary angiography as well as in the carotid artery (intima-media-thickness) and peripheral vessels (ankle brachial index). Association analysis of genetic and metabolic markers with atherosclerotic burden will be performed to identify novel factors of disposition to atherosclerotic vascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients assigned to coronary angiography

Exclusion Criteria:

* Cancer
* Acute myocardial infarction
* Inability to give informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients assigned to coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Thiery, MD PhD, Principal Investigator — University of Leipzig
Locations (2):
- Germany (2):
  - University of Leipzig, Institute of Laboratory Medicine, Clinical Chemistry and Molecular Diagnostics, Leipzig
  - University of Leipzig, Heart Center, Department of Cardiology, Leipzig

REFERENCES:
- [Derived] Teren A, Vogel A, Beutner F, Gielen S, Burkhardt R, Scholz M, Thiery J, Ceglarek U. Relationship between fermented dairy consumption, circulating short-chain acylcarnitines and angiographic severity of coronary artery disease. Nutr Metab Cardiovasc Dis. 2020 Sep 24;30(10):1662-1672. doi: 10.1016/j.numecd.2020.05.031. Epub 2020 Jun 8. PMID 32684363
- [Derived] Jacobi T, Massier L, Kloting N, Horn K, Schuch A, Ahnert P, Engel C, Loffler M, Burkhardt R, Thiery J, Tonjes A, Stumvoll M, Bluher M, Doxiadis I, Scholz M, Kovacs P. HLA Class II Allele Analyses Implicate Common Genetic Components in Type 1 and Non-Insulin-Treated Type 2 Diabetes. J Clin Endocrinol Metab. 2020 Mar 1;105(3):dgaa027. doi: 10.1210/clinem/dgaa027. PMID 31974565
- [Derived] Pott J, Schlegel V, Teren A, Horn K, Kirsten H, Bluecher C, Kratzsch J, Loeffler M, Thiery J, Burkhardt R, Scholz M. Genetic Regulation of PCSK9 (Proprotein Convertase Subtilisin/Kexin Type 9) Plasma Levels and Its Impact on Atherosclerotic Vascular Disease Phenotypes. Circ Genom Precis Med. 2018 May;11(5):e001992. doi: 10.1161/CIRCGEN.117.001992. PMID 29748315
- [Derived] Weissgerber A, Scholz M, Teren A, Sandri M, Teupser D, Gielen S, Thiery J, Schuler G, Beutner F. The value of noncoronary atherosclerosis for identifying coronary artery disease: results of the Leipzig LIFE Heart Study. Clin Res Cardiol. 2016 Feb;105(2):172-81. doi: 10.1007/s00392-015-0900-x. Epub 2015 Sep 11. PMID 26362881
- [Derived] Beutner F, Teupser D, Gielen S, Holdt LM, Scholz M, Boudriot E, Schuler G, Thiery J. Rationale and design of the Leipzig (LIFE) Heart Study: phenotyping and cardiovascular characteristics of patients with coronary artery disease. PLoS One. 2011;6(12):e29070. doi: 10.1371/journal.pone.0029070. Epub 2011 Dec 22. PMID 22216169
- See also: University Hospital Leipzig, Institute of Laboratory Medicine, Clinical Chemistry and Molecular Diagnostics — http://ilm.uniklinikum-leipzig.de/index.php?lang=en